CLINICAL TRIAL: NCT05209204
Title: Anterior Chamber Angle Examination in Angle Closure Suspect Patients
Status: Completed | Type: Observational
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mohamed Salah, MD, Minia University
Other Study IDs: AC angle angle closure suspect
Record Dates: First submitted 2022-01-07; First posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Glaucoma
Keywords: Angle closure; ASOCT
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 40 pateint glucoma suspect: ASOCT
  Interventions: Diagnostic Test: ASOCT; Diagnostic Test: Pentacam

INTERVENTIONS:
Diagnostic Test: ASOCT — Anterior segment imaging using RTVue XR 100 Avanti OCT platform (Optovue Inc.,Fairmont, CA).
Diagnostic Test: Pentacam — Anterior segment imaging using Oculus Pentacam HR (Oculus Optikgeräte, Wetzlar, Germany).

SUMMARY:
The aim of this study is to detect PACG suspects using both AS OCT and Scheimpflug imaging.

DETAILED DESCRIPTION:
Glaucoma is a form of progressive optic neuropathy and is one of the leading causes of preventable blindness worldwide. The average life span is increasing leading to more individuals developing glaucoma as well as having the disease longer, which makes early detection and management very important.[1] Glaucoma is characterized by loss of retinal ganglion cells (RGCs) recognized as optic nerve head (ONH) changes, corresponding visual field (VF) defects and retinal nerve fiber layer (RNFL) loss. At least 40% of RGCs are lost before the VFs show a defect, hence the emphasis on early diagnosis in the stage of glaucoma suspect.[2] There are two types of glaucoma suspect: Primary Open angle and primary angle closure suspect.(3) Primary angle-closure (PAC) suspects can be detected by the following: the trabecular meshwork can only be seen in 180º or less of anterior chamber angle (AC) by gonioscopy, the intraocular pressure(IOP) remains within normal limits and no structural damage to the optic nerve is present.[4] Time domain Optical coherence tomography (TD-OCT) was initially designed to image the posterior segment and retina, but its capability to generate cross-sectional images of internal biological structures without contacting the ocular surface was quickly adapted to visualize the anterior segment and cornea.[5].

Spectral domain anterior segment OCT (SD-OCT) technology allow visualizing the anterior chamber angle of the eye with high speed and high resolution. Spectral-domain OCT(SD OCT) instruments working at 840 nm can reliably identify fine angle structures such as Schwalbe's line.(6) Scheimpflug imaging also offers non-contact imaging of the anterior segment. Although Scheimpflug photography cannot fully visualize the entire angle, the software available on the Pentacam system (Oculus Optikgeräte, Wetzlar, Germany) provides extrapolated measurements of the anterior chamber volume (ACV), which have shown promise in screening for narrow angles.(7)

ELIGIBILITY:
Inclusion Criteria:

* Hyperopes. 2-Shallow AC. 3-With gonioscopy carried out under dim-light conditions without indentation ,with the eye in primary position there is inability to visualize ≤ 180° of the posterior trabecular meshwork (TM) in the absence of peripheral anterior 4-IOP ≤ 21 as measured by tonometry. 5-Normal visual field on static automated perimetry (SAP) testing. 5-Normal optic nerve head (ONH) appearance on fundus biomicroscopy. 6-Family history of primary angle closure disease.

Exclusion Criteria:

* 1-Eyes with significant corneal opacity that can impare signal strings of any of the used imaging modalities.

  2-Eyes wih history of intraocular surgery (e.g. cataract surgery ,retinal detachment surgery).

  3-Eyes with history of laser procedures (e.g.laser peripheral iridotomy). 4-Eyes with anterior segment pathology as iridocyclitis or angle disgenesis 5. Eyes with history of trauma. 6- Eyes with findings suggestive of 2dry cause of glaucoma (e.g. iris or angle neovascularization, any iris or corneal abnormalities, dilated episcleral vessels ).

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Residents of Minia Governorate diagnosed with SLE with renal affection and without renal affection.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Anterior segment parameters as measured by AS-OCT: | 3 months
  Anterior chamber depth (ACD)..
Anterior segment parameters as measured by Oculus Pentacam: | 3 months
  Anterior chamber angle (ACA).
Anterior segment parameters by ASOCT | 3 months
  Angle opening distance at 750 µm (AOD750).
Anterior segment parameters by OCT | 3 months
  Anterior chamber angle (ACA).
Pentacam parameters | 3 months
  Anterior chamber volume (ACV).
Pentacam parameters by Oculus Pentacam: | 3 months
  Anterior chamber depth (ACD).

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Salah, Principal Investigator — Minia University Hospital
Locations (1):
- Minia University hospital, Minya, Egypt